CLINICAL TRIAL: NCT02663479
Title: Proprietary Lipid-Lowering Nutraceutical Supplement in the Management of Hypertension
Brief Title: Nutraceutical Supplement in the Management of Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thorne HealthTech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TruCardia-002
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Cardiopressin (Experimental): A 5 capsule proprietary blend of herbal extracts and nutrients
  Interventions: Dietary Supplement: Cardiopressin
- Placebo (Placebo Comparator): A 5 capsule placebo matched in color and size to the Experimental supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cardiopressin
  Arms: Cardiopressin
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a proprietary nutraceutical supplement in capsule form over 4 months in treating blood pressure in a group of chronic hypertensive subjects that are not receiving any pharmaceutical anti-hypertensive agents or other nutraceutical supplements.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with chronic hypertension: Blood pressure at study entry must be greater than or equal to systolic blood pressure of 140 mm Hg but less than 180 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg but less than 105 mm Hg
* Subjects are not taking any prescription anti-hypertensive drugs.
* Subjects must be off all nutraceutical supplements for at least 30 days prior to entry into the study.

Exclusion Criteria

* Myocardial infarction, PTCA , stent, CABG within 5 years, known clinical CHD or clinical angina.
* History of cerebrovascular accident (CVA).
* Creatinine over 2.5 mg/dL.
* Known allergy or sensitivity to any components of the study blood pressure supplement.
* Chronic liver disease with AST, ALT, alkaline phosphatase over 1.5 x normal lab values.
* Known cancer within 2 years.
* Clinical congestive heart failure ( systolic or diastolic CHF)
* Pregnant and nursing women and women.
* Women of child bearing age not on approved contraception control.
* Type 1 and Type 2 diabetes mellitus on medications.
* If the study subjects develop BP over 180 mm Hg systolic or 110 mm Hg diastolic during the study, they will be discontinued from the study and the investigator will immediately start rescue drug therapy for BP control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 4 months
  Reduction in systolic and diastolic blood pressure as measured by office readings and 24 hour ABM ( ambulatory blood pressure monitor)

SECONDARY OUTCOMES:
Endothelial Function | 4 months
  Measured via Endopat
Small arterial compliance | 4 months
  Measured via computerized arterial pulse wave analysis (CAPWA)
Large arterial compliance | 4 months
  Measured via computerized arterial pulse wave analysis (CAPWA)
Central arterial blood pressure | 4 months
  Measured via computerized arterial pulse wave analysis (CAPWA)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Houston, MD, MS, MSc, Principal Investigator — Hypertension Institute; Bodi Zhang, MD, MPH, PhD, Principal Investigator — Thorne Research
Locations (1):
- Hypertension Institute of Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No